CLINICAL TRIAL: NCT00183404
Title: Long-Term Olanzapine Treatment in Children With Autism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01MH073524 (NIH); R01MH073524 (NIH); DDTR B2-NDA (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Autism
Keywords: Drug Treatment; Child; Olanzapine
MeSH Terms: conditions — Autistic Disorder | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Olanzapine (Experimental): Participants will take open olanzapine for up to 20 additional weeks after phase 1.
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Olanzapine tablets, dosed once or twice per day, dosage 2.5 to 20 mg per day
  Other Names: Open Olanzapine

SUMMARY:
This study will determine the short- and long-term safety and effectiveness of the drug olanzapine (Zyprexa®) for reducing symptoms of autism in children.

DETAILED DESCRIPTION:
Autism is a serious childhood disorder that can significantly impair functioning and development. Educational and psychosocial programs are standard treatments for autistic children, but drug therapy is often needed as well. Haloperidol is the drug most commonly prescribed for symptoms of autism. However, long-term administration of haloperidol has been associated with adverse effects such as blurred vision, constipation, and nausea. The investigation of alternative drug treatments is necessary. This study will determine whether the antipsychotic drug olanzapine may be a safe and effective alternative to haloperidol for treating symptoms of autism in children.

This study will last 36 weeks and will comprise 2 phases. In Phase I, participants will be randomly assigned to receive either olanzapine or placebo for 12 weeks. Participants who do not respond to treatment will complete their participation in the study. Participants who respond to their assigned Phase I treatment will continue onto Phase II. All Phase II participants will receive olanzapine daily for 6 months. Self-report scales and checklists will be used to assess participants after each phase; these measures will be completed by participants and their parents.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism
* Parent or guardian willing to provide informed consent

Exclusion Criteria:

* Uncontrolled seizure disorder
* Medical illness other than autism affecting the whole body
* Obesity
* History of psychosis
* Impairment of voluntary movement
* History of olanzapine treatment

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2004-09; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Children's Psychiatric Rating Scale | Measured monthly throughout the study

SECONDARY OUTCOMES:
Aberrant Behavior Checklist | Measured monthly throughout the study
Clinical Global Impressions | Measured monthly throughout the study
Treatment Emergent Symptoms Scale | Measured monthly throughout the study
Olanzapine Untoward Effects Checklist | Measured monthly throughout the study
Abnormal Involuntary Movement Scale | Measured monthly throughout the study
Neurological Rating Scale | Measured monthly throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Richard P. Malone, MD, Principal Investigator — Drexel University College of Medicine
Locations (1):
- Drexel University College of Medicine at Friends Hospital, Philadelphia, Pennsylvania, United States